CLINICAL TRIAL: NCT06256575
Title: Treatment of Digital Ulcers in Systemic Sclerosis With Diosmin: A Randomized, Double-blind, Placebo-controlled Multi-centre Pilot Study
Brief Title: Study of Diosmin for the Treatment of Digital Ulcers in Systemic Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVDUS-01
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-05

CONDITIONS: Scleroderma, Systemic; Digital Ulcer
Keywords: SSc; Digital Ulcers; Sclerosis; Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers; Sclerosis; Scleroderma, Diffuse | interventions — Diosmin

STUDY DESIGN:
Intervention Model Description: This is a parallel study of two (2) arms in which participants receive different interventions. Participants are randomized and assigned to the treatment or placebo arm at the beginning of the trial. They continue in that arm throughout the length of the trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects de-identified, all study staff blinded, all product labeled with number assignment, randomization performed by computer, number assignment conveyed to blinded study staff via computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Vasculera 630 mg, tablet, two (2) times per day for eight (8) weeks
  Interventions: Combination Product: Diosmin
- Placebo (Placebo Comparator): Cornstarch, one (1) capsule, two (2) times per day for eight (8)
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Diosmin — A medical food of diosmin and alka4-complex
  Other Names: Vasculera
  Arms: Active
Other: Placebo — Corn starch one (1) capsule twice daily
  Arms: Placebo

SUMMARY:
This study is performed to consider the safety and healing ability of diosmin in patients with systemic sclerosis (scleroderma) and open sores on their fingers (digital ulcers). Two (2) out of three (3) participants will receive active product. The participants will have four (4) visits over eight (8) weeks. Physical exams and photos will be performed. A variety of questions will be asked describing level of pain and lifestyle changes.

DETAILED DESCRIPTION:
This study is performed to consider the safety and healing ability of diosmin in patients with systemic sclerosis (scleroderma) and open sores on their fingers (digital ulcers). The study will include 21-45 participants randomly given active product or inactive product (placebo). Two (2) out of every three (3) participants enrolled will receive active product. The participants will have four (4) visits over eight (8) weeks. At each visit physical exams and photos will be performed. Each person will also be asked a variety of questions describing level of pain and any changes to their lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic sclerosis (scleroderma)
* At least one "active" digital ulcer
* Medication for systemic sclerosis unchanged for 30 days

Exclusion Criteria:

* Infection or gangrene in ulcer
* Citrus allergy
* Unstable heart, kidney, or liver disease
* Active infection of any type
* Current cancer treatment or uncured cancer
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Number (%) of healed baseline ulcers | Screening, Day 1, Day 28, Day 56
  Number (%) of healed baseline ulcers and change in net ulcer burden

SECONDARY OUTCOMES:
Safety - number of adverse events | Screening, Day 1, Day 28, Day 56
  The number of product related adverse events experienced

CONTACTS AND LOCATIONS:
Overall Officials: Lukban, Study Director — Primus Pharmaceuticals
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Dalhousie University, Halifax, Nova Scotia
  - Saint Joseph Health Care Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Health System, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: Primus director of clinical research will review requests submitted via email.